CLINICAL TRIAL: NCT04085094
Title: Gender Differences in Renal Disease Progression: an Analysis of Potential Mechanisms Using Modern Radiological Techniques
Brief Title: Gender Differences in Renal Functioning and Disease
Acronym: GenderBOLD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Gregoire Wuerzner; MD, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: 2016-01971
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Chronic Renal Failure; Healthy Controls
Keywords: BOLD-MRI; Contrast-enhanced ultrasound (CEUS); Salt storage; Perfusion index; Resistance index; Renal functional reserve; Renal oxygenation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — myotrophin; Diet, Sodium-Restricted; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of blood samples (all), urine (all) and sweat in some.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1. Healthy and pre-menopausal women without CKD: A total of 45 healthy and pre-menopausal women (<50 years old) will be recruited. Thirty of them are not on oral anticonception; 15 will be examined at each visit during their follicular phase, 15 during their luteal phase. Fifteen are on oral contraception.
  Three visits will take place:
  * V1: after 5 days of a high salt diet (adding 6g of salt/day on top of regular diet), patients will undergo renal ultrasound (Doppler and CEUS), renal functional MRI (BOLD and phase contrast) and Na23 muscle and skin MRI.
  * V2: after 5 days of low salt diet (dietary instructions), the same exams mentioned above will be repeated
  * V3: renal CEUS will be performed before and after an oral protein load (1g/kg) or after SL nitroglycerin (0.2mg).
  The day before each visit, a 24h urine collection will be performed in order to measure renal salt excretion.
  Interventions: Dietary Supplement: high-salt diet (V1) and low salt diet (V2); Diagnostic Test: Contrast-enhanced ultrasound (CEUS); Diagnostic Test: functional MRI; Other: Pilocarpine test
- 2. Pre-menopausal women with CKD: A total of 30 women with CKD will be recruited and undergo the same visits as outlined above
  Interventions: Dietary Supplement: high-salt diet (V1) and low salt diet (V2); Diagnostic Test: Contrast-enhanced ultrasound (CEUS); Diagnostic Test: functional MRI
- 3. Post-menopausal women without CKD: Fifteen post-menopausal women will undergo the same exams as outlined above
  Interventions: Dietary Supplement: high-salt diet (V1) and low salt diet (V2); Diagnostic Test: Contrast-enhanced ultrasound (CEUS); Diagnostic Test: functional MRI
- 4. Healthy men: A total of thirty age-and sex-matched men (15 below and 15 above 50 years old) will undergo the same exams as above.
  Interventions: Dietary Supplement: high-salt diet (V1) and low salt diet (V2); Diagnostic Test: Contrast-enhanced ultrasound (CEUS); Diagnostic Test: functional MRI; Other: Pilocarpine test
- 5.Men with CKD: Fifteen men with CKD will undergo the same exams as outlined above
  Interventions: Diagnostic Test: Contrast-enhanced ultrasound (CEUS); Diagnostic Test: functional MRI

INTERVENTIONS:
Dietary Supplement: high-salt diet (V1) and low salt diet (V2) — Before the first visit, the participant will follow a five-day high salt diet (addition of 6g/day of salt to their regular diet followed at home). Before the second visit (V2), the participant will follow for five days a low-salt diet, according to dietary instructions followed provided during the screening visit.
  Groups: 1. Healthy and pre-menopausal women without CKD; 2. Pre-menopausal women with CKD; 3. Post-menopausal women without CKD; 4. Healthy men
Diagnostic Test: Contrast-enhanced ultrasound (CEUS) — Renal ultrasound with use of a contrast product (SonoVue®), perfusion rate 0.015ml/kg/min. Four destruction-reperfusion sequences are performed in order to measure the Perfusion Index (PI) of the renal cortex.
Diagnostic Test: functional MRI — Measurement of renal oxygenation with the Blood Oxygenation Level Dependant-MRI technique (BOLD-MRI) on Siemens Prisma 3T scanner before and 15minutes after 0.03mg/kg of IV furosemide. Assessment of the amount of salt stored in the skin and muscles with the 23Na MRI technique.
Other: Pilocarpine test — Assessment of sweat salt and potassium concentrations in healthy volunteers according to slat intake. Two electrodes are placed on the forearm. The electric current between the two electrodes will induce perspiration which will be collected with the Macroduct system.
  Groups: 1. Healthy and pre-menopausal women without CKD; 4. Healthy men

SUMMARY:
The purpose of the GenderBOLD study is to shed light on the mechanisms responsible for women's lower susceptibility to developing and progressing chronic renal disease, using modern imaging techniques, and applying different diets. The investigators postulate that oxygenation and renal perfusion are better conserved and change less in women than in men in different dietary situations (high salt-low salt), possibly because they are able to store excess salt in their skin and muscles. The investigators postulate that these differences are independent of their menstrual cycle. Finally, the investigators will analyze the renal functional reserve and changes in renal perfusion through an oral protein load and after sublingual nitroglycerin to assess whether potential différences exist between genders.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) affects about 10% of the adult population in Switzerland.

Despite decades of research, the mechanisms involved in the development and progression of CKD remain unclear, and there is a lack of preventative therapies. Women are relatively protected against CKD, but this topic has been little studied.

The kidney is very sensitive to hypoxia and its chronic oxygen depravation is the final step in the pathogenesis of CKD. A special MRI application, called BOLD-MRI, has the ability to measure renal tissue oxygenation in humans. In a recent BOLD-MRI study, the investigators demonstrated that cortical oxygenation is significantly higher in women than in men, which may explain women's lower susceptibility to declining renal function. However, whether this is true under different dietary conditions (high salt-low salt), and whether renal oxygenation changes throughout the menstrual cycle is unknown and will be assessed in this study.

Renal oxygenation depends on its perfusion. Renal micro-perfusion can be measured with contrast-enhanced ultrasound (CEUS) and is expressed as PI (perfusion index). CEUS is a recent imaging technique that combines conventional ultrasound with the administration of a microbubble contrast agent (a lipid or albumin-enveloped gas compound). The microbubbles are inert and eliminated by pulmonary and hepatic systems within one hour of administration. They are not nephrotoxic and have no major side effects. Whether there are differences in renal perfusion as measured with CEUS between men and women with and without CKD will be also assessed in this study.

Oxygenation of the kidneys does not only depend on their perfusion, but also on their consumption, mainly related to tubular active sodium transport. Thus, their oxygenation is lower in the case of a high salt diet compared to a low salt diet. This has been proven in men, but not in women.

Recently, another MRI technique called 23Na MRI was used to measure the amount of salt stored in the skin and muscles. It is possible that the cutaneous and muscular capacity of storing salt according to dietary salt intake is lower in men, but this has not, at present, been examined.

ELIGIBILITY:
Inclusion/exclusion Criteria:

Inclusion criteria for healthy pre-menopausal women:

* Age ≥ 18 years old and <50 years old.
* No drugs (psychoactive substances used for non-medical purposes) /medicine.
* Blood pressure <135/85mmHg.
* Renal function (eGFR >90ml/min/1.73m2) and absence of albuminuria.
* Regular menstrual cycle.
* No pregnancy.
* Understanding and signature of the informed consent.

Inclusion criteria for pre-menopausal women with a chronic renal failure:

* Age ≥ 18 years old and <50 years old.
* Possibility to stop the treatment during the day of the study.
* Reduced renal function (eGFR 15-60 ml/min/1.73m2) or eGFR 60-90 ml/min/1.73m2 with the presence of albuminuria >300 mg/j.
* Understanding and signature of the informed consent.

Inclusion criteria for post-menopausal women:

* Age ≥ 50 years old.
* Absence of menstruation.
* No drugs consumption.
* No medicine, or possibility to stop it two days before the study.
* Blood pressure <135/85mmHg.
* Renal function (eGFR >90ml/min/1.73m2) and absence of albuminuria.
* Understanding and signature of the informed consent.

Inclusion criteria for men:

* Age ≥ 18 years old, but matched with the age of pre- aor post-menopausal women
* No drugs consumption.
* No medicine, or possibility to stop it two days before the study.
* Blood pressure <135/85mmHg.
* Renal function (eGFR >90ml/min/1.73m2) and absence of albuminuria.
* Understanding and signature of the informed consent.

Exclusion criteria for all:

* Contra-indication for Magnetic Resonance Imaging (Pacemaker, implanted metallic device, claustrophobia,..)
* Known allergy to one of the study compounds (furosemide, Sonovue).

Exclusion criteria for persons with chronic renal failure:

* Autosomal dominant polycystic kidney disease.
* Ingestion of corticosteroids or other immunosuppressants.
* Volume overload or heart failure.
* eGFR < 15ml/min/1.73m2 or dialysis.

Exclusion criteria for men and women receiving sublingual nitroglycerin:

* Hypersensitivity to nitrous derivatives or to one of the excipients present in the composition.
* History of heart disease (ischemic heart disease, valve and/or rhythmic).
* Low blood pressure (systolic blood pressure <100mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is characterized by several groups which contain only men or only women.
Study Population: Healthy volunteers will be recruited by way of advertisement at CHUV. Patients with CKD will be recruited via the ambulatory nephrology consultation.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Change in renal microperfusion according to dietary salt intake in healthy and CKD | 1 month (5 days high salt- two weeks wash out- 5 days low salt)
  Renal perfusion is measured with the contrast-enhanced ultrasound (CEUS)
Change in renal oxygenation after salty/unsalted diets in women compared to men | 1 month
  Renal oxygenation is measured by Blood Oxygen Level Dependent (BOLD-IRM)
Change in skin and muscle storage of sodium according to salt intake | 1 month
  Changes in cutaneous and muscle sodium storage measured by 23Na-MRI
Change in renal perfusion measured with CEUS after SL nitroglycerine | before-5 minutes after NTG
  Renal perfusion is measured with the contrast-enhanced ultrasound (CEUS)

CONTACTS AND LOCATIONS:
Overall Officials: Menno Pruijm, PD MD, Principal Investigator — CHUV
Locations (1):
- CHUV, nephrology service, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No